CLINICAL TRIAL: NCT04459247
Title: Short Term, High Dose Vitamin D Supplementation for COVID-19 Disease: Double Blind, Controlled, Study
Brief Title: Short Term, High Dose Vitamin D Supplementation for COVID-19
Acronym: SHADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121/20
Record Dates: First submitted 2020-07-03; First posted 2020-07-07 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: COVID

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Vitamin D high dose
  Interventions: Drug: Vit D
- Control arm (No Intervention): No Vitamin D supplementation

INTERVENTIONS:
Drug: Vit D — Oral liquid formulation of 60000 IU
  Arms: Intervention

SUMMARY:
Coronavirus-2019 (COVID-19) caused by severe acute respiratory syndrome-associated coronavirus-2 (SARS-CoV-2) has affected the lives of millions of individuals globally and severely strained the medical community. Pre-symptomatic and asymptomatic SARS-CoV-2 positive individuals far outnumber the symptomatic ones or those with severe disease. The transmission potential of SARS CoV-2 is potentially greator than earlier viral outbreaks of SARS-CoV and MERS-CoV. Identification of asymptomatic carriers of SARS-CoV-2 infection is paramount to contain viral infection because of high transmission potential Routine measures of social distancing, personal hand hygiene and limited outdoor contact activities have shown benefits to limit corona virus infection. However, the role of vitamin D in SARS-CoV-2 infection is not explored despite the knowledge of an immunomodulatory role and protective effect of vitamin D against viral infections. It has been found that mortality from COVID-19 is more in countries with vitamin D deficiency.

The role of therapeutic vitamin D supplementation in asymptomatic individuals with vitamin-D deficiency and COVID-19 is not known. Immune-modulatory effect of vitamin D is likely to be observed at 25(OH)D levels which are considered higher than that required for normal bone metabolism.An earlier SARS-CoV-2 negativity may have significant public health benefits in limiting the spread of the disease. Therefore, we hypothesise that high dose vitamin D supplementation in patients with COVID-19 and vitamin D deficiency may lead to SARS-CoV-2 negativity in greater proportions of patients associated with decrease in serological markers of inflammation.

DETAILED DESCRIPTION:
The role of therapeutic vitamin D supplementation in asymptomatic individuals with vitamin-D deficiency and COVID-19 is not known. Immune-modulatory effect of vitamin D is likely to be observed at 25(OH)D levels which are considered higher than that required for normal bone metabolism.[6] An earlier SARS-CoV-2 negativity may have significant public health benefits in limiting the spread of the disease. Therefore, we hypothesise that high dose vitamin D supplementation in patients with COVID-19 and vitamin D deficiency may lead to SARS-CoV-2 negativity in greater proportions of patients associated with decrease in serological markers of inflammation.

Methods: Consecutive individuals with SARS-CoV-2 infection who were mildly symptomatic or asymptomatic with or without co-morbidities (hypertension, diabetes mellitus, chronic obstructive airway disease, chronic liver disease) admitted to tertiary care hospital in north India were invited for the study. A written consent was obtained from all patients included in the study and protocol was approved by the Institute Ethics Committee.

Patients with vitamin D deficiency defined as 25 (OH)D level<20 ng/ml were randomized to receive daily 60,000IU of cholecalciferol (5 ml oral solution in nano droplet form) for seven days in the "intervention arm" or to receive a single dose of 60,000 IU vitamin D supplementation at admission in the "control arm". Patients unable to take oral supplementation like those requiring invasive ventilation were excluded. Subsequently, 25(OH)D levels were assessed at day 7 and a weekly supplementation of 60,000IU provided to those with 25(OH)D >50 ng/ml or continued on daily vitamin D 60,000 IU supplementation for another seven days in participants with 25 (OH)D<50ng/ml (day-14) in the intervention arm. No vitamin D supplementation was provided in the control arm other than the initial dose at hospital admission.

25 (OH)D, serum calcium, phosphorus, fibrinogen , d-dimer, C-reactive protein, procalcitonin, renal and liver function tests were performed periodically up till day-21 or virus negativity, whichever occurred earlier. Oro-pharyngeal swabs were obtained for SARS-CoV-2 RNA detection at day-5, 7, 10, 14, 18 and 21 and detection was performed by real-time polymerase chain reaction (RT-PCR), CFX-96 IVD, Bio-Rad. 25 (OH)D was analysed by electrochemiluminescence immunoassay (ECLIA) (Roche Cobas E 801 Analyzer; Roche Diagnostics), using the kit supplied by the same manufacturer (Elecsys Total Vitamin D, version 2.0). Serum calcium (N, 8.5-10.2 mg/dl) and C-reactive protein (N, 0-5 mg/l) were processed by ECLIA method using Roche Cobas 8000, Roche Diagnostics. D dimer (N, 0-240 ng/ml) & fibrinogen (N, 2-4g/l) were analyzed using Stago Compact/ Stago STA R model, Diagnostica Stago, Inc, USA respectively.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 RNA positive Asymptomatic individuals

Exclusion Criteria:

* Uncontrolled Diabetes Uncontrolled Hypertension Chronic Liver Disease Chronic obstructive Pulmonary disease Requiring Invasive Ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Virus negativity | 21 days
  SARS-CoV-2 RNA negative

SECONDARY OUTCOMES:
Inflammatory Marker | 21 days
  Change in fibrinogenLevels
Inflammatory Marker 2 | 21 days
  Change in D-Dimer Levels

CONTACTS AND LOCATIONS:
Locations (1):
- Deptt of Endocrinology, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stroehlein JK, Wallqvist J, Iannizzi C, Mikolajewska A, Metzendorf MI, Benstoem C, Meybohm P, Becker M, Skoetz N, Stegemann M, Piechotta V. Vitamin D supplementation for the treatment of COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 24;5(5):CD015043. doi: 10.1002/14651858.CD015043. PMID 34029377
- [Derived] Rastogi A, Bhansali A, Khare N, Suri V, Yaddanapudi N, Sachdeva N, Puri GD, Malhotra P. Short term, high-dose vitamin D supplementation for COVID-19 disease: a randomised, placebo-controlled, study (SHADE study). Postgrad Med J. 2022 Feb;98(1156):87-90. doi: 10.1136/postgradmedj-2020-139065. Epub 2020 Nov 12. PMID 33184146